CLINICAL TRIAL: NCT01978509
Title: The Affect of Low-Volume Bowel Preparation for Hospitalized Patients Colonoscopies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Francisco C. Ramirez, M.D., MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 13-003983
Record Dates: First submitted 2013-09-23; First posted 2013-11-07 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Colonoscopy
Keywords: Colonoscopy
MeSH Terms: interventions — MoviPrep; Golytely

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low volume prep (Prepopik) (Active Comparator): Low volume prep for colonoscopy (Prepopik)
  Interventions: Drug: Low volume prep (Prepopik)
- Moderate volume prep (Moviprep) (Active Comparator): Moderate volume prep for colonoscopy (Moviprep)
  Interventions: Drug: Moderate volume prep (Moviprep)
- High volume prep (Golytely) (Active Comparator): High volume prep for colonoscopy (Golytely)
  Interventions: Drug: High volume prep (Golytely)

INTERVENTIONS:
Drug: Low volume prep (Prepopik) — Hospitalized patients will be randomized to receive either large volume bowel preparation (Golytely), moderate volume bowel prep (Moviprep) or low volume bowel preparation (Prepopik) in a split dose manner for bowel cleansing prior to colonoscopy.
  Other Names: Prepopik
  Arms: Low volume prep (Prepopik)
Drug: Moderate volume prep (Moviprep) — Hospitalized patients will be randomized to receive either large volume bowel preparation (Golytely), moderate volume bowel prep (Moviprep) or low volume bowel preparation (Prepopik) in a split dose manner for bowel cleansing prior to colonoscopy.
  Other Names: Moviprep
  Arms: Moderate volume prep (Moviprep)
Drug: High volume prep (Golytely) — Hospitalized patients will be randomized to receive either large volume bowel preparation (Golytely), moderate volume bowel prep (Moviprep) or low volume bowel preparation (Prepopik) in a split dose manner for bowel cleansing prior to colonoscopy.
  Other Names: Golytely
  Arms: High volume prep (Golytely)

SUMMARY:
The purpose of this study is to compare the efficacy of a low-volume bowel preparation versus a high-volume bowel preparation for bowel cleansing on hospitalized patients undergoing colonoscopies.

ELIGIBILITY:
Inclusion criteria:

1. Inpatient colonoscopy
2. Age 18 years and older
3. Able to give consent
4. Split dose colonoscopies for all patients

Exclusion criteria:

1. Unable to give consent
2. Pregnant or lactating women
3. Renal impairment (GFR <30)
4. Ileus
5. Ascites
6. Toxic megacolon
7. Gastrointestinal obstruction
8. Allergy to study drugs
9. Toxic colitis
10. Not able to split the dose of bowel preparations to be used
11. Contraindication to bowel preparation
12. Risk for aspiration
13. Risk of severe cardiac arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Ramirez, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Derived] Hernandez PV, Horsley-Silva JL, Snyder DL, Baffy N, Atia M, Koepke L, Buras MR, Lim ES, Ruff K, Umar SB, Islam S, Ramirez FC. Effect of bowel preparation volume in inpatient colonoscopy. Results of a prospective, randomized, comparative pilot study. BMC Gastroenterol. 2020 Jul 13;20(1):227. doi: 10.1186/s12876-020-01373-1. PMID 32660521
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Volume Prep (Prepopik) | Moderate Volume Prep (Moviprep) | High Volume Prep (Golytely)
Started | 10 | 13 | 9
Completed | 8 | 8 | 9
Not Completed | 2 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Volume Prep (Prepopik) | Moderate Volume Prep (Moviprep) | High Volume Prep (Golytely) | Total
Number analyzed (Participants) | 10 | 13 | 9 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (17.54) | 56.13 (19.08) | 70.78 (12.33) | 63.66 (17.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 3 | 12
  Male | 8 | 6 | 6 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 13 | 9 | 32

OUTCOME MEASURES:

1. Primary Outcome: Bowel Cleansing
Description: Measured using the total Boston Bowel Prep Score (BBPS) obtained by adding scores from each segment for a range of minimum 0 = very poor and maximum 9 = excellent.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Volume Prep (Prepopik) | Moderate Volume Prep (Moviprep) | High Volume Prep (Golytely)
Number analyzed (Participants) | 8 | 8 | 9
score on a scale | 7.4 (1.62) | 6.9 (1.55) | 7.0 (1.41)
Statistical Analysis 1: Comparison: Low Volume Prep (Prepopik) vs Moderate Volume Prep (Moviprep) vs High Volume Prep (Golytely); Test type: Superiority; p = 0.70, ANOVA

2. Secondary Outcome: Cancellation or Delay of Procedure Due to Poor Bowel Preparation
Description: To assess the rate of delayed and or cancellation of procedure due to inadequate bowel preparation
Time Frame: 24 hours
Population: Study was terminated due to lack of enrollment and data not collected.
Arm/Group | Low Volume Prep (Prepopik) | Moderate Volume Prep (Moviprep) | High Volume Prep (Golytely)
Number analyzed (Participants) | 0 | 0 | 0

3. Other Pre Specified Outcome: Patient Tolerance
Description: Percentage of participants self-reporting finishing the bowel preparation
Time Frame: 24 hours
Measure: Number; unit: percentage of participants
Arm/Group | Low Volume Prep (Prepopik) | Moderate Volume Prep (Moviprep) | High Volume Prep (Golytely)
Number analyzed (Participants) | 8 | 8 | 9
percentage of participants | 100 | 75 | 77.8

4. Other Pre Specified Outcome: Cecal Intubation
Description: Assess the success of cecal intubation rate between three bowel preparations.
Time Frame: 24 hours
Population: Study was terminated due to lack of enrollment and data not collected.
Arm/Group | Low Volume Prep (Prepopik) | Moderate Volume Prep (Moviprep) | High Volume Prep (Golytely)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected on all participants from study enrollment to study completion, approximately 24 hours. Adverse events were collected throughout the duration of the entire study, approximately 7 years.
Arm/Group | Low Volume Prep (Prepopik) | Moderate Volume Prep (Moviprep) | High Volume Prep (Golytely)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/13 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/13 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/13 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT01978509/Prot_000.pdf